CLINICAL TRIAL: NCT04569032
Title: A Dual-cohort, Open-label, Phase 2 Study of Brentuximab Vedotin and CHP (A+CHP) in the Frontline Treatment of Subjects With Peripheral T-cell Lymphoma (PTCL) With Less Than 10% CD30 Expression
Brief Title: A Study of Brentuximab Vedotin and CHP in Frontline Treatment of PTCL With Less Than 10% CD30 Expression
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Seagen, a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Organization: Seagen Inc. (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SGN35-032
Record Dates: First submitted 2020-09-23; First posted 2020-09-29 (Actual); Results first posted 2025-05-15 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Peripheral T-cell Lymphoma
Keywords: CD30-positive; CD30-negative; Seattle Genetics
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — Brentuximab Vedotin; Cyclophosphamide; Doxorubicin; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CD30-negative Cohort (Experimental): Participants with CD30 expression level < 1%
  Interventions: Drug: brentuximab vedotin; Drug: cyclophosphamide; Drug: doxorubicin; Drug: prednisone
- CD30-positive Cohort (Experimental): Participants with CD30 expression level ≥1% to < 10%
  Interventions: Drug: brentuximab vedotin; Drug: cyclophosphamide; Drug: doxorubicin; Drug: prednisone

INTERVENTIONS:
Drug: brentuximab vedotin — 1.8 mg/kg administered intravenously (IV; into the vein) on Day 1 of each 21 -day cycle
  Other Names: ADCETRIS
Drug: cyclophosphamide — 750 mg/m^2 administered intravenously (IV; into the vein) on Day 1 of each 21 -day cycle
Drug: doxorubicin — 50 mg/m^2 administered intravenously (IV; into the vein) on Day 1 of each 21 -day cycle
Drug: prednisone — 100 mg daily administered orally on Days 1-5 of each cycle

SUMMARY:
This clinical trial will study brentuximab vedotin with CHP to find out if the drugs work for people who have certain types of peripheral T-cell lymphoma (PTCL). It will also find out what side effects occur when brentuximab vedotin and CHP are used together. A side effect is anything the drugs do besides treating cancer. CHP is a type of chemotherapy that uses three drugs (cyclophosphamide, doxorubicin, and prednisone). CHP is approved by the FDA to treat certain types of PTCL.

ELIGIBILITY:
Inclusion Criteria

* Newly diagnosed PTCL, excluding systemic anaplastic large cell lymphoma (sALCL), per the Revised European-American Lymphoma World Health Organization (WHO) 2016 classification
* The following non-sALCL PTCL subtypes are eligible:

  * PTCL - not otherwise specified (PTCL-NOS)
  * Angioimmunoblastic T-cell lymphoma (AITL)
  * Adult T-cell leukemia/lymphoma (ATLL; acute and lymphoma types only, must be positive for human T cell leukemia virus 1)
  * Enteropathy-associated T-cell lymphoma (EATL)
  * Hepatosplenic T-cell lymphoma
  * Monomorphic epitheliotropic intestinal T-cell lymphoma (MEITCL)
  * Indolent T-cell lymphoproliferative disorder (T-LPD) of the gastrointestinal (GI) tract
  * Follicular T-cell lymphoma
  * Nodal peripheral T-cell lymphoma with T-follicular helper (TFH) phenotype
* CD30 expression <10% by local assessment in tumor containing lymph node or other extranodal soft tissue biopsy
* Fluorodeoxyglucose (FDG)-avid disease by PET and measurable disease of at least 1.5 cm by CT, as assessed by the site radiologist
* An Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2

Exclusion Criteria

* Current diagnosis of any of the following:

  * sALCL
  * Primary cutaneous T-cell lymphoproliferative disorders and lymphomas
  * Mycosis fungoides (MF), including transformed MF
* History of another primary invasive cancer, hematologic malignancy, or myelodysplastic syndrome that has not been in remission for at least 3 years. Exceptions are malignancies with a negligible risk of metastasis or death (e.g., 5-year OS ≥90%), such as carcinoma in situ of the cervix, non-melanoma skin carcinoma, localized prostate cancer, ductal carcinoma in situ, or Stage I uterine cancer.
* History of progressive multifocal leukoencephalopathy (PML).
* Cerebral/meningeal disease related to the underlying malignancy.
* Prior treatment with brentuximab vedotin or doxorubicin.
* Baseline peripheral neuropathy Grade 2 or higher (per the NCI CTCAE, Version 4.03) or subjects with the demyelinating form of Charcot-Marie-Tooth syndrome.
* Left ventricular ejection fraction less than 45% or symptomatic cardiac disease (including symptomatic ventricular dysfunction, symptomatic coronary artery disease, and symptomatic arrhythmias), or myocardial infarction within the past 6 months, or previous treatment with complete cumulative dose of >300 mg/m2 of doxorubicin.
* Any uncontrolled Grade 3 or higher (per the National Cancer Institute's Common Terminology Criteria for Adverse Events, NCI CTCAE Version 4.03) viral, bacterial, or fungal infection within 2 weeks prior to the first dose of study drug. Routine antimicrobial prophylaxis is permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2020-11-12 (Actual); Primary Completion 2024-05-09 (Actual); Study Completion 2025-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (63):
- United States (43):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Stanford Cancer Center, Stanford, California
  - Stanford Hospital and Clinics, Investigational Drug Services, Stanford, California
  - Rocky Mountain Cancer centers, LLP, Aurora, Colorado
  - Rocky Mountain Cancer centers, LLP, Boulder, Colorado
  - Rocky Mountain Cancer centers, LLP, Colorado Springs, Colorado
  - Rocky Mountain Cancer centers, LLP, Denver, Colorado
  - Rocky Mountain Cancer centers, LLP, Lakewood, Colorado
  - Rocky Mountain Cancer centers, LLP, Littleton, Colorado
  - Rocky Mountain Cancer centers, LLP, Lone Tree, Colorado
  - Rocky Mountain Cancer centers, LLP, Longmont, Colorado
  - Rocky Mountain Cancer centers, LLP, Pueblo, Colorado
  - Rocky Mountain Cancer centers, LLP, Thornton, Colorado
  - Tulane Cancer Center, New Orleans, Louisiana
  - Tulane Medical Center, New Orleans, Louisiana
  - Memorial Sloan Kettering Cancer Center David H. Koch Center for Cancer Care, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Oncology_Hematology Care Clincal Trials,LLC, Cincinnati, Ohio
  - Cleveland Clinic taussig Cancer Center Investigational Pharmacy, Cleveland, Ohio
  - Cleveland Clinic, The, Cleveland, Ohio
  - Oncology_Hematology Care Clincal Trials,LLC, Fairfield, Ohio
  - Texas Oncology - Central/South Texas, Austin, Texas
  - Texas Oncology - Central South (Balcones Dr), Austin, Texas
  - Texas Oncology - Central South (James Casey), Austin, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - US Oncology Investigational Products Center (IPC), Irving, Texas
  - US Oncology Investigational Products Center(IPC), Irving, Texas
  - US Oncology lnvestigational Products Center (IPC), Irving, Texas
  - Texas Oncology-Northeast Texas, Longview, Texas
  - Texas Oncology-Northeast Texas, Palestine, Texas
  - Texas Oncology-Northeast Texas, Paris, Texas
  - Texas Oncology-Northeast Texas, Tyler, Texas
  - Virginia Oncology Associates, Chesapeake, Virginia
  - Virginia Oncology Associates, Hampton, Virginia
  - Virginia Oncology Associates, Newport News, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - VCU Massey Cancer Center-Radiation Oncology, Richmond, Virginia
  - VCU Medical Center -InPatient, Richmond, Virginia
  - VCU Medical Center Critical Care Hospital, Richmond, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - VCU at Stony Point, Richmond, Virginia
  - Massey Cancer Center Clinical & Translational Research Lab, Richmond, Virginia
  - Virginia Oncology Associates, Virginia Beach, Virginia
- France (3):
  - CHU Grenoble Alpes, Tranche, Auvergne-Rhône-Alpes
  - Hopital Emile Muller, Mulhouse
  - Höpital Haut Levéque - CHU Bordeaux Service d'hématologie clinique et thérapie cellulaire, Pessac
- Italy (6):
  - Azienda Ospedaliero Universitaria di Bologna - IRCCS, Bologna, Emilia-Romagna
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Lombardy
  - Fondazione Irccs San Matteo, Pavia, Lombardy
  - IRCCS Ospedale Policlinico San Martino, Genova, Other
  - Fondazione del Piemonte per l'Oncologia (FPO) - IRCCS Candiolo - Oncologia Medica, Candiolo, Turin
  - Azienda Ospedaliera Universitaria Integrata Verona Policlinico G.B. Rossi, Verona
- Spain (6):
  - IEC Trials, Hospital La Milagrosa., Madrid, Other
  - Hospital Universitario De La Paz, Madrid, Other
  - Cetir Centre Medic, Barcelona
  - Hospital Duran I Reynals - Institut Catala d'Oncologia, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Clinico Universitario de Salamanca, Salamanca
- United Kingdom (5):
  - Oxford University Hospitals, Headington, Other
  - UCLH Hospitals, London
  - Hammersmith Hospital, London
  - MACMILLIAN Cancer Centre, London
  - The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who had newly diagnosed non-systemic anaplastic large cell lymphoma (sALCL) peripheral T-cell lymphoma (PTCL) with < 10% CD30 expression, were enrolled to receive A+CHP treatment (brentuximab vedotin, cyclophosphamide, doxorubicin, and prednisone). Enrollment was based on CD30 expression per local laboratory assessment. Analysis of efficacy outcome measures was based on CD30 expression per central laboratory assessment.
Pre-assignment Details: Results reported are based on the primary completion date (PCD) of the study; data for only those secondary outcome measures are reported for which analyses were complete at PCD. Remaining outcome measures would be reported upon completion of their analyses at study completion.
Groups:
- CD30 <1% [Local Laboratory Assessment]: Participants with <1% CD30 expression (per local laboratory assessment) received A+CHP treatment in 21-day cycle. Brentuximab vedotin as 1.8 milligrams per kilogram (mg/kg) intravenously (IV) on Day 1 of each 21-day cycle, Cyclophosphamide 750 milligram per square meter (mg/m^2) IV on Day 1 of each 21-day cycle, Doxorubicin 50 mg/m^2 IV on Day 1 of each 21-day cycle, Prednisone 100 mg orally on Days 1-5 of each 21-day cycle.
- CD30 1% to <10% [Local Laboratory Assessment]: Participants with 1% to <10% CD30 expression (per local laboratory assessment) received A+CHP treatment in 21-day cycle. Brentuximab vedotin as 1.8 mg/kg IV on Day 1 of each 21-day cycle, Cyclophosphamide 750 mg/m^2 IV on Day 1 of each 21-day cycle, Doxorubicin 50 mg/m^2 IV on Day 1 of each 21-day cycle, Prednisone 100 mg orally on Days 1-5 of each 21-day cycle.
Period: Overall Study
Arm/Group | CD30 <1% [Local Laboratory Assessment] | CD30 1% to <10% [Local Laboratory Assessment]
Started (Based on Local Laboratory Assessment) | 34 | 48
Completed | 0 | 0
Not Completed | 34 | 48
Not completed — Death | 10 | 13
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — In long term follow up | 22 | 34

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CD30 <1% [Local Laboratory Assessment] | CD30 1% to <10% [Local Laboratory Assessment] | Total
Number analyzed (Participants) | 34 | 48 | 82
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.2 (11.3) | 61.0 (11.0) | 60.7 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 26 | 36
  Male | 24 | 22 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 10 | 19
  Not Hispanic or Latino | 22 | 34 | 56
  Unknown or Not Reported | 3 | 4 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 4 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 26 | 37 | 63
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) Per Blinded Independent Central Review (BICR) by Revised Response Criteria for Malignant Lymphoma Criteria (Cheson 2007) by Central CD30 Assessment
Description: ORR was defined as the percentage of participants with complete response (CR) or partial response (PR) following the completion of study treatment (at end of treatment [EOT]). CR and PR per Cheson 2007: CR was defined as complete disappearance of all detectable clinical evidence of disease and disease-related symptoms if present before therapy and PR was defined as at least a 50% decrease in sum of the product of the diameters (SPD) of up to six of the largest dominant nodes or nodal masses.
Time Frame: At EOT or the first assessment after the last dose of study treatment (prior to long term follow-up or initiation of subsequent anti-cancer therapies); up to 41.91 months
Population: Full analysis set (FAS) included all participants who received any amount of brentuximab vedotin or any component of cyclophosphamide, doxorubicin, and prednisone (CHP). Analyses as planned was based on the participants classified based on central laboratory assessment for CD30 expression.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- CD30 <1% [Central Laboratory Assessment]: Participants with <1% CD30 expression (per central laboratory assessment) received A+CHP treatment in 21-day cycle. Brentuximab vedotin as 1.8 mg/kg IV on Day 1 of each 21-day cycle. Cyclophosphamide 750 mg/m^2 IV on Day 1 of each 21-day cycle, Doxorubicin 50 mg/m^2 IV on Day 1 of each 21-day cycle, Prednisone 100 mg orally on Days 1-5 of each 21-day cycle.
- CD30 1% to <10% [Central Laboratory Assessment]: Participants with 1% to <10% CD30 expression (per central laboratory assessment) received A+CHP treatment in 21-day cycle. Brentuximab vedotin as 1.8 mg/kg IV on Day 1 of each 21-day cycle. Cyclophosphamide 750 mg/m^2 IV on Day 1 of each 21-day cycle, Doxorubicin 50 mg/m^2 IV on Day 1 of each 21-day cycle, Prednisone 100 mg orally on Days 1-5 of each 21-day cycle.
Arm/Group | CD30 <1% [Central Laboratory Assessment] | CD30 1% to <10% [Central Laboratory Assessment]
Number analyzed (Participants) | 23 | 31
Percentage of participants | 61 [38.5 to 80.3] | 81 [62.5 to 92.5]

2. Secondary Outcome: Complete Response (CR) Rate Per BICR (Cheson 2007) by Central CD30 Assessment
Description: CR rate was defined as the percentage of participants with CR following the completion of study treatment (at EOT). CR as per Cheson 2007: CR was defined as complete disappearance of all detectable clinical evidence of disease and disease-related symptoms if present before therapy.
Time Frame: as for outcome 1
Population: FAS included all participants who received any amount of brentuximab vedotin or any component of CHP. Analyses as planned was based on the participants classified based on central laboratory assessment for CD30 expression.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | CD30 <1% [Central Laboratory Assessment] | CD30 1% to <10% [Central Laboratory Assessment]
Number analyzed (Participants) | 23 | 31
Percentage of participants | 52 [30.6 to 73.2] | 71 [52.0 to 85.8]

3. Secondary Outcome: Progression Free Survival (PFS) Per BICR (Cheson 2007) by Central CD30 Assessment
Description: PFS was defined as the time from start of study treatment to the first documentation of objective tumor progression or to death due to any cause, whichever came first. Kaplan-Meier method was used for analysis. PFS data was censored on the date of the last radiological assessment of measured lesions documenting absence of PD for participants without objective tumor progression and were still on study at the time of an analysis, were given antitumor treatment other than the study treatment or stem cell transplant (included donor lymphocyte infusion) or were removed from study prior to documentation of objective tumor progression. Participants who lacked an evaluation of tumor response after their first dose had their event time censored at 1 day.
Time Frame: From the first dose of study treatment to first documentation of objective tumor progression or death due to any cause or censoring, whichever came first (approximately 61.7 months)
Reporting Status: Not Posted, anticipated posting 2025-12

4. Secondary Outcome: Overall Survival (OS) by Central CD30 Assessment
Description: OS was defined as the time from first dose to death due to any cause. Participant not known to have died by the end of study follow-up, observation of OS was censored on the date the participants were last known to be alive (i.e., date of last contact). Participants who lacked data beyond the day of first dose had their survival time censored on the date of first dose (i.e., OS duration of 1 day). Kaplan-Meier method was used for analysis.
Time Frame: From the first dose of study treatment until death or censoring date, whichever came first (approximately 61.7 months)
Reporting Status: Not Posted, anticipated posting 2025-12

5. Secondary Outcome: Duration of Response (DOR) Per BICR (Cheson 2007) by Central CD30 Assessment
Description: DOR was defined as the time from the first documentation of objective tumor response (CR or PR) to the first documentation of tumor progression (per Cheson 2007) or death, whichever came first. Participants without progression or death were censored. DOR was only calculated for the subset of participants achieving a CR or PR. CR and PR per Cheson 2007: CR was defined as complete disappearance of all detectable clinical evidence of disease and disease-related symptoms if present before therapy and PR was defined as at least a 50% decrease in sum of the product of the diameters (SPD) of up to six of the largest dominant nodes or nodal masses. Kaplan-Meier method was used for analysis.
Time Frame: From the first documented CR or PR until the first documentation of tumor progression, death or censoring date, whichever came first (up to 61.7 months)
Reporting Status: Not Posted, anticipated posting 2025-12

6. Secondary Outcome: ORR Per BICR by Modified Lugano Criteria (Cheson 2014) by Central CD30 Assessment
Description: ORR was defined as the percentage of participants with CR or PR following the completion of study treatment (at EOT) according to the modified Lugano criteria (Cheson 2014). Complete response was defined as complete disappearance of radiologic evidence of disease and PR was defined as at least a 50% decrease in SPD of up to six of the largest dominant nodes or nodal masses.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | CD30 <1% [Central Laboratory Assessment] | CD30 1% to <10% [Central Laboratory Assessment]
Number analyzed (Participants) | 23 | 31
Percentage of participants | 57 [34.5 to 76.8] | 77 [58.9 to 90.4]

7. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Treatment Emergent Serious Adverse Events (TESAEs) and Treatment Related Adverse Events by Local CD30 Assessment
Description: An adverse event was any untoward medical occurrence in a participant or clinical investigational participant administered a medicinal product and which did not necessarily have a causal relationship with this treatment. An adverse event was classified as a serious adverse event (SAE) if it met one of the following criteria: fatal, life threatening, hospitalization, disabling/incapacitating, congenital anomaly or birth defect or any medically significant event. TEAEs were events if they were newly occurring or worsen following study treatment. TESAE is any SAE that met treatment emergent definition. Treatment related AEs were which had evidence to suggest a causal relationship between the drugs and the adverse event, such as: an event that was uncommon and known to be strongly associated with drug exposure, an event that was not commonly associated with drug exposure but was otherwise uncommon in the population exposed to the drug. AEs included both SAEs and all non-SAEs.
Time Frame: From first dose of the study treatment (Day 1) up to 30-37 days after the last dose of study treatment (approximately up to 6.6 months)
Population: FAS included all participants who received any amount of brentuximab vedotin or any component of CHP.
Measure: Count of Participants; unit: Participants
Arm/Group | CD30 <1% [Local Laboratory Assessment] | CD30 1% to <10% [Local Laboratory Assessment]
Number analyzed (Participants) | 34 | 48
Participants
  TEAEs | 32 | 46
  TESAEs | 15 | 16
  Treatment related TEAEs | 25 | 40

8. Secondary Outcome: Number of Participants With Treatment Emergent Laboratory Abnormalities as Per Worst Post Baseline Grading, by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.03 by Local CD30 Assessment
Description: Any Abnormal laboratory tests(Decreased values of hemoglobin,leukocytes,lymphocytes,neutrophils, platelets, calcium corrected for albumin,glomerular filtration rate estimated, glucose, phosphate, potassium,albumin,sodium and increased values of calcium corrected for albumin,creatinine, potassium, glucose, alanine aminotransferase, alkaline phosphatase, aspartate aminotransferase, total Bilirubin, urate) that worsen from baseline were considered clinically significant by investigator.Abnormal test were recorded as AE if associated with accompanying symptoms,required additional diagnostic testing or medical/surgical intervention,study dosing change,study discontinuation,significant additional concomitant drug treatment,other therapy.As perNCI CTCAE grade(G)1:mild(asymptomatic or mild symptoms,clinical,diagnostic observations,no intervention),G2:moderate(minimal, local,noninvasive intervention),G3:severe,medically significant,G4:life-threatening,urgent intervention,G5:death related to AE
Time Frame: as for outcome 7
Population: FAS included all participants who received any amount of brentuximab vedotin or any component of CHP. Here, "Overall Number of Participants Analyzed" were participants evaluable for this outcome measure however all participants reported under "Overall Number of Participants Analyzed' contributed data to table but may not have evaluable data for every row. Here, "Number Analyzed" signifies participants evaluable for the specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | CD30 <1% [Local Laboratory Assessment] | CD30 1% to <10% [Local Laboratory Assessment]
Number analyzed (Participants) | 34 | 48
Participants
  Hemoglobin decreased: Grade 1+2: number analyzed (Participants) | 33 | 47
  Hemoglobin decreased: Grade 1+2 | 19 | 34
  Hemoglobin decreased: Grade 3: number analyzed (Participants) | 33 | 47
  Hemoglobin decreased: Grade 3 | 3 | 1
  Leukocytes decreased: Grade 1+2: number analyzed (Participants) | 33 | 47
  Leukocytes decreased: Grade 1+2 | 13 | 23
  Leukocytes decreased: Grade 3: number analyzed (Participants) | 33 | 47
  Leukocytes decreased: Grade 3 | 4 | 5
  Leukocytes decreased: Grade 4: number analyzed (Participants) | 33 | 47
  Leukocytes decreased: Grade 4 | 0 | 1
  Lymphocytes decreased: Grade 1+2: number analyzed (Participants) | 33 | 47
  Lymphocytes decreased: Grade 1+2 | 10 | 15
  Lymphocytes decreased: Grade 3: number analyzed (Participants) | 33 | 47
  Lymphocytes decreased: Grade 3 | 15 | 21
  Lymphocytes decreased: Grade 4: number analyzed (Participants) | 33 | 47
  Lymphocytes decreased: Grade 4 | 1 | 4
  Neutrophils decreased: Grade 1+2: number analyzed (Participants) | 33 | 47
  Neutrophils decreased: Grade 1+2 | 3 | 12
  Neutrophils decreased: Grade 3: number analyzed (Participants) | 33 | 47
  Neutrophils decreased: Grade 3 | 4 | 3
  Neutrophils decreased: Grade 4: number analyzed (Participants) | 33 | 47
  Neutrophils decreased: Grade 4 | 1 | 3
  Platelets decreased: Grade 1+2: number analyzed (Participants) | 33 | 47
  Platelets decreased: Grade 1+2 | 6 | 10
  Platelets decreased: Grade 4: number analyzed (Participants) | 33 | 47
  Platelets decreased: Grade 4 | 0 | 1
  Calcium Corrected for Albumin increased: Grade 1+2: number analyzed (Participants) | 32 | 46
  Calcium Corrected for Albumin increased: Grade 1+2 | 3 | 1
  Creatinine increased: Grade 1+2: number analyzed (Participants) | 33 | 47
  Creatinine increased: Grade 1+2 | 19 | 30
  Glomerular Filtration Rate, Estimated decreased: Grade 1+2: number analyzed (Participants) | 18 | 31
  Glomerular Filtration Rate, Estimated decreased: Grade 1+2 | 2 | 4
  Glucose decreased: Grade 1+2: number analyzed (Participants) | 33 | 47
  Glucose decreased: Grade 1+2 | 1 | 5
  Glucose increased: Grade 1+2: number analyzed (Participants) | 33 | 47
  Glucose increased: Grade 1+2 | 15 | 21
  Glucose increased: Grade 3: number analyzed (Participants) | 33 | 47
  Glucose increased: Grade 3 | 3 | 0
  Glucose increased: Grade 4: number analyzed (Participants) | 33 | 47
  Glucose increased: Grade 4 | 0 | 1
  Phosphate decreased: Grade 1+2: number analyzed (Participants) | 31 | 46
  Phosphate decreased: Grade 1+2 | 1 | 1
  Phosphate decreased: Grade 3: number analyzed (Participants) | 31 | 46
  Phosphate decreased: Grade 3 | 0 | 4
  Potassium decreased: Grade 1+2: number analyzed (Participants) | 33 | 47
  Potassium decreased: Grade 1+2 | 2 | 5
  Potassium decreased: Grade 3: number analyzed (Participants) | 33 | 47
  Potassium decreased: Grade 3 | 1 | 1
  Potassium decreased: Grade 4: number analyzed (Participants) | 33 | 47
  Potassium decreased: Grade 4 | 0 | 1
  Alanine Aminotransferase increased: Grade 1+2: number analyzed (Participants) | 33 | 47
  Alanine Aminotransferase increased: Grade 1+2 | 6 | 17
  Albumin decreased: Grade 1+2: number analyzed (Participants) | 32 | 46
  Albumin decreased: Grade 1+2 | 3 | 8
  Alkaline Phosphatase increased: Grade 1+2: number analyzed (Participants) | 33 | 43
  Alkaline Phosphatase increased: Grade 1+2 | 2 | 11
  Alkaline Phosphatase increased: Grade 3: number analyzed (Participants) | 33 | 43
  Alkaline Phosphatase increased: Grade 3 | 2 | 0
  Aspartate Aminotransferase increased: Grade 1+2: number analyzed (Participants) | 33 | 47
  Aspartate Aminotransferase increased: Grade 1+2 | 8 | 15
  Aspartate Aminotransferase increased: Grade 3: number analyzed (Participants) | 33 | 47
  Aspartate Aminotransferase increased: Grade 3 | 0 | 1
  Calcium Corrected for Albumin decreased: Grade 1+2: number analyzed (Participants) | 32 | 46
  Calcium Corrected for Albumin decreased: Grade 1+2 | 2 | 2
  Potassium increased: Grade 1+2: number analyzed (Participants) | 33 | 47
  Potassium increased: Grade 1+2 | 2 | 4
  Potassium increased: Grade 3: number analyzed (Participants) | 33 | 47
  Potassium increased: Grade 3 | 1 | 0
  Sodium decreased: Grade 1+2: number analyzed (Participants) | 33 | 47
  Sodium decreased: Grade 1+2 | 8 | 6
  Sodium decreased: Grade 3: number analyzed (Participants) | 33 | 47
  Sodium decreased: Grade 3 | 1 | 3
  Sodium increased: Grade 1+2: number analyzed (Participants) | 33 | 47
  Sodium increased: Grade 1+2 | 0 | 2
  Total Bilirubin increased: Grade 1+2: number analyzed (Participants) | 33 | 47
  Total Bilirubin increased: Grade 1+2 | 1 | 1
  Urate increased: Grade 3: number analyzed (Participants) | 33 | 47
  Urate increased: Grade 3 | 4 | 6
  Urate increased: Grade 4: number analyzed (Participants) | 33 | 47
  Urate increased: Grade 4 | 2 | 0

ADVERSE EVENTS:
Time Frame: Adverse events: From first dose of the study treatment (Day 1) maximum up to 30-37 days after the last dose of study treatment (approximately up to 6.6 months). All-cause mortality: throughout the study (up to 41 months)
Description: Same event may appear as both non-serious adverse event and serious adverse event (SAE); however, are presented as distinct events. Event may be categorized as serious in 1 participant and non-serious in another or may have experienced both SAE and non-SAE. Results are reported based on participants classified per local laboratory assessment for CD30 expression.
Arm/Group | CD30 <1% [Local Laboratory Assessment] | CD30 1% to <10% [Local Laboratory Assessment]
All-Cause Mortality (participants affected / at risk) | 11/34 | 13/48
Serious Adverse Events (participants affected / at risk) | 15/34 | 16/48
Other Adverse Events (participants affected / at risk) | 31/34 | 43/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CD30 <1% [Local Laboratory Assessment] (N=34) | CD30 1% to <10% [Local Laboratory Assessment] (N=48)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 6 (7) | 9 (15)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Malabsorption (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 4 (4) | 1 (1)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Herpes simplex reactivation (Infections and infestations) | 0 (0) | 1 (1)
Pseudomonal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection pseudomonal (Infections and infestations) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Cutaneous T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bell's palsy (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1)
Cognitive disorder (Nervous system disorders) | 0 (0) | 1 (1)
Nervous system disorder (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CD30 <1% [Local Laboratory Assessment] (N=34) | CD30 1% to <10% [Local Laboratory Assessment] (N=48)
Anaemia (Blood and lymphatic system disorders) | 7 (7) | 15 (18)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 5 (6)
Neutropenia (Blood and lymphatic system disorders) | 4 (4) | 12 (19)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 4 (4)
Constipation (Gastrointestinal disorders) | 3 (3) | 7 (7)
Diarrhoea (Gastrointestinal disorders) | 6 (9) | 19 (25)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 3 (3)
Nausea (Gastrointestinal disorders) | 8 (11) | 14 (21)
Stomatitis (Gastrointestinal disorders) | 1 (3) | 6 (6)
Vomiting (Gastrointestinal disorders) | 4 (4) | 7 (8)
Asthenia (General disorders) | 5 (7) | 3 (3)
Fatigue (General disorders) | 4 (4) | 7 (7)
Oedema peripheral (General disorders) | 5 (5) | 6 (7)
Pyrexia (General disorders) | 2 (2) | 8 (19)
COVID-19 (Infections and infestations) | 2 (2) | 4 (5)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 4 (4)
Neutrophil count decreased (Investigations) | 2 (2) | 1 (1)
Weight decreased (Investigations) | 4 (4) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 4 (4)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 7 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Dizziness (Nervous system disorders) | 4 (4) | 0 (0)
Dysgeusia (Nervous system disorders) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 4 (5) | 2 (2)
Paraesthesia (Nervous system disorders) | 3 (3) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 3 (3) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 11 (12) | 16 (18)
Insomnia (Psychiatric disorders) | 2 (2) | 4 (4)
Pollakiuria (Renal and urinary disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 7 (7)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 6 (6)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 1 (1)
Embolism (Vascular disorders) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 3 (4) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-03-10): https://cdn.clinicaltrials.gov/large-docs/32/NCT04569032/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-16): https://cdn.clinicaltrials.gov/large-docs/32/NCT04569032/SAP_001.pdf